CLINICAL TRIAL: NCT02353078
Title: The Effect of Sucralfate Slurry on Dilated Intercellular Spaces, Tight Junctions, Mucosal Impedance and Mucosal Activity in Patients With Eosinophilic Esophagitis
Brief Title: The Effect of Sucralfate Slurry in Patients With Eosinophilic Esophagitis
Acronym: EoE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David A. Katzka, David A. Katzka, MD, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-008661
Record Dates: First submitted 2015-01-26; First posted 2015-02-02 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis (EOE)
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Sucralfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sucralfate (Experimental): This is a pilot study in which 6 patients with active EoE defined by consensus criteria (ref) who have undergone recent endoscopy will be administered sucralfate slurry 1 gram four times daily for four weeks following which repeat endoscopy with esophageal biopsies will be performed. Patients will be those who had not had medical treatment for EoE or those who have not responded to proton pump inhibitors.
  Interventions: Drug: Sucralfate
- Intraluminal Impedance (Experimental): This procedure involves passing a mucosal impedance probe through the endoscope and gently placing the tip of the probe on the esophageal mucosa. Measurements will be made at 2,5,10 and 15 cm above the gastroesophageal junction. There is no increased risk to the procedure and it adds approximately 2 minutes to the procedure.
  Interventions: Procedure: Intraluminal Impedance; Device: Intraluminal Impedance

INTERVENTIONS:
Drug: Sucralfate — Sucralfate slurry 1 gram four times daily for four weeks
  Other Names: Carafate
  Arms: Sucralfate
Procedure: Intraluminal Impedance — During the initial endoscopy, esophageal mucosal impedance will also be measured. This procedure involves passing a mucosal impedance probe through the endoscope and gently placing the tip of the probe on the esophageal mucosa. Measurements will be made at 2,5,10 and 15 cm above the gastroesophageal junction. There is no increased risk to the procedure and it adds approximately 2 minutes to the procedure.
  Other Names: Mucosal Impedance
  Arms: Intraluminal Impedance
Device: Intraluminal Impedance — The mucosal impedance probe is a 2.13 mm catheter (tiny tube), called an Intraluminal Impedance, will be passed through the channel of the standard endoscope. There is no increased risk to the procedure and it adds approximately 2 minutes to the procedure.
  Other Names: Mucosal Impedance
  Arms: Intraluminal Impedance

SUMMARY:
Could Sucralfate be a non-steriodal treatment option for patients with Eosinophilic esophagitis?

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EoE) is a Th2 type allergy mediated disease that is characterized by dense esophageal eosinophilia in patients with chronic esophageal symptoms. One of the mechanisms of eosinophilic esophagitis is exposure of food antigens to antigen recognition cells in the esophageal mucosa that initiates a chronic allergy-based inflammatory response [1, 2]. It is believed that this exposure is facilitated through dilation of the intercellular spaces (DIS) between esophageal epithelial cells (termed spongiosis). This is substantiated by several studies which have demonstrated that: first, DIS is commonly found in biopsies from patients with active EoE and reverses with steroid therapy [3]; second, DIS correlates to physiologic demonstration of increased esophageal epithelial permeability as shown through transepithelial small molecule flux in mucosal biopsies appraised in Ussing chambers [4], and third, DIS is associated with decreased expression of specific epithelial tight junction proteins such as filaggrin [3]. Thus, a suggested sequence of events in EoE that leads to allergen initiated inflammation includes down regulation of tight junction proteins, dilation of intercellular spaces in the surface epithelium followed by increased permeability and facilitated exposure to food antigens.

Of the present therapies available, topical steroids and in a subset of EoE patients, proton pump inhibitors may improve epithelial permeability. Unfortunately, in the case of proton pump inhibitors, there is early data suggesting that their therapeutic benefit is not sustained. With the use of steroids, there are fears of what the long term side effects of continued use of swallowed steroids might be. The other alternative treatment, diet exclusion therapy is difficult to tailor to the patient and impractical for most adult patients. As a result, alternative treatments are need for EoE.

Sucralfate is a medication that was developed for the treatment of acid-peptic diseases. It's mechanism of action in healing lesions such as gastroduodenal mucosal ulceration still remains unclear but has been described as a "cytoprotective" agent. Several mechanisms have been suggested to be responsible for this protection. These include: binding to and protection of exposed eroded areas, increased prostaglandin production, improved vascular flow, and increased mucus production. This compound has also been shown to augment potential difference in gastric mucosa suggesting a decreased in ion flow. The investigators have shown in measuring mucosal impedance in EoE, this may be related to closure of intercellular spaces which could make this an attractive therapy for eosinophilic esophagitis. Furthermore, the side effect profile of sucralfate is excellent with little systemic absorption. Sucralfate is a category (B) medication, safe for females of child bearing years.

ELIGIBILITY:
Inclusion criteria:

• Patients between the ages of 18 and 80 with eosinophilic esophagitis diagnosed by a combination of compatible symptoms, endoscopic findings, histology, and lack of response to proton pump inhibitors.

Exclusion criteria:

* Medical conditions such as severe heart or lung disease that preclude safe performance of endoscopy
* Pregnant and lactating females will be excluded
* Diabetic patients will be excluded as episodes of hyperglycemia have been reported
* Patient with chronic renal failure/on dialysis will be excluded
* Patients with conditions known to be associated with esophageal eosinophilia, including Crohn's disease, Churg-Strauss, achalasia, and hypereosinophilic syndrome
* Inability to read due to: Blindness, cognitive dysfunction, or English language illiteracy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The Effectiveness of Sucralfate treatment in patient's with EoE | 4 weeks
  • The effect treatment is defined by 50%, 3 of the 6 patients having less < 15 eosinophilia per high power field by in the pathology at the time of follow up endoscopic biopsies.

SECONDARY OUTCOMES:
Measuring Mucosal impedance | 4 weeks
  Mucosal impedance reflects the ability of electric current to flow between two sensors while in contact with the epithelium. An increase in current flow is presumably due to an increase in ions and water crossing the membrane, which are good conductors of electricity. Through this technique an overall measure of "leakiness" of the esophageal epithelium is obtained. This increased permeability may reflect epithelial destruction as in erosive esophagitis and Eosinophilic esophagitis. The investigators will measure the mucosal impedance at the baseline during the upper endoscopy and at the follow up endoscopy. Comparing these measurement to the eosinophilic count on pathology at baseline and followup.

CONTACTS AND LOCATIONS:
Overall Officials: David Katzka, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States